CLINICAL TRIAL: NCT00004038
Title: Pilot Study of p53 Intralesional Gene Therapy With Chemotherapy in Breast Cancer
Brief Title: Gene Therapy Plus Chemotherapy in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02273; FCCC-97009; NCI-T97-0042; CDR0000066480 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-12-10; First posted 2004-05-20 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2001-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — advexin; Drug Therapy

ARMS (1):
- Arm I (Experimental): Patients undergo biopsy of one of their skin nodules prior to any treatment. Patients receive the Ad-p53 gene therapy in one nodule and injection of a second nodule with Dulbecco's phosphate buffered saline. The next day, patients begin chemotherapy, which may be given weekly and continues every 21-28 days for up to 6 courses. On day 3, patients return for biopsy of injected nodules. Biopsies are only performed during the first course. Patients may receive further injections of the Ad-p53 gene with subsequent courses of chemotherapy, for up to six courses.
  Interventions: Biological: Ad5CMV-p53 gene; Drug: chemotherapy

INTERVENTIONS:
Biological: Ad5CMV-p53 gene
Drug: chemotherapy

SUMMARY:
Phase I trial to study the effectiveness of gene therapy plus chemotherapy in treating patients who have breast cancer. Inserting the p53 gene into a person's cancer cells may improve the body's ability to fight cancer or make the cancer more sensitive to chemotherapy. Combining chemotherapy with gene therapy may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the effect of adenovirus p53 (Ad-p53) on chemotherapy-induced apoptosis in lesions in patients with breast cancer.

II. Determine p53 protein expression following intralesional injections of Ad-p53 by immunohistochemistry and reverse transcriptase polymerase chain reaction in this patient population.

III. Determine the time course and magnitude of the development of a humoral antibody response to the adenoviral vector in this patient population.

IV. Determine the ability of transfected p53 to upregulate downstream signals important in G1 arrest by assaying for WAF1 mRNA and apoptosis in this patient population.

V. Determine the toxicities and side effects of intralesional injections of Ad-p53 given in combination with standard chemotherapy in patients with cutaneous and subcutaneous metastatic breast cancer amenable to injections and biopsies.

VI. Determine if there is an increase in apoptosis induced by Ad-53 compared to baseline in this patient population.

OUTLINE:

Patients undergo biopsy of one of their skin nodules prior to any treatment. Patients receive the Ad-p53 gene therapy in one nodule and injection of a second nodule with Dulbecco's phosphate buffered saline. The next day, patients begin chemotherapy, which may be given weekly and continues every 21-28 days for up to 6 courses. On day 3, patients return for biopsy of injected nodules. Biopsies are only performed during the first course. Patients may receive further injections of the Ad-p53 gene with subsequent courses of chemotherapy, for up to six courses.

Patients are followed monthly for 4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed epithelial breast cancer
* At least 3 cutaneous or subcutaneous lesions required
* Measurable disease that includes, but is not limited to, cutaneous or subcutaneous metastases

PATIENT CHARACTERISTICS:

* Age: Over 18
* Performance status: ECOG 0-2
* Absolute granulocyte count at least 1,500/mm3
* Hemoglobin greater than 8 g/dL
* Platelet count greater than 100,000/mm3
* Bilirubin less than 2 mg/dL
* PT/PTT within normal range
* SGOT/SGPT less than 2 times upper limit of normal
* Creatinine less than 1.8 mg/dL
* Not pregnant
* Fertile patients must use effective contraception during and for 3 months after therapy

PRIOR CONCURRENT THERAPY:

* Concurrent cytotoxic chemotherapy allowed, if stable and responding
* At least 4 weeks since prior chemotherapy, if starting a new regimen
* At least 4 weeks since radiotherapy
* Prior adjuvant radiotherapy to the chest wall allowed
* At least 6 months since radiotherapy to lesions that are to be injected
* Recovered from prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1999-01; Primary Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States